CLINICAL TRIAL: NCT02722096
Title: Creation of Arteriovenous Ante-brachial Fistula Under Axillary Block Versus Local Anesthesia : Impact on Early Complications
Acronym: FAV ss ALR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013.829
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Kidney Failure, Chronic
Keywords: arteriovenous fistula; regional anesthesia; local anesthesia; early complication
MeSH Terms: conditions — Kidney Failure, Chronic; Arteriovenous Fistula | interventions — Ropivacaine; Lidocaine; Anesthesia, Local

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Axillary block anesthesia (Experimental): Axillary brachial plexus block anesthesia (with Ropivacaine and Lidocaine) will be performed by anesthetist 30 to 45 minutes before surgery
  Interventions: Drug: Axillary block anesthesia with Ropivacaine and Lidocaine
- Local anesthesia (Active Comparator): Local subcutaneous infiltration of Ropivacaine and Lidocaine will be performed by anesthetist at the beginning of surgery
  Interventions: Drug: Local anesthesia with Ropivacaine and Lidocaine

INTERVENTIONS:
Drug: Axillary block anesthesia with Ropivacaine and Lidocaine — Axillary brachial plexus block anesthesia with injection of Ropivacaine and Lidocaine will be performed by anesthetist 30 to 45 minutes before surgery
  Arms: Axillary block anesthesia
Drug: Local anesthesia with Ropivacaine and Lidocaine — Local subcutaneous infiltration of Ropivacaine and Lidocaine will be performed by anesthetist at the beginning of surgery
  Arms: Local anesthesia

SUMMARY:
Recommended by the KDOQI vascular access guidelines, antebrachial arteriovenous fistula is the best primary vascular access for hemodialysis in patients with end stage renal disease. The primary complications are common, of the order of 10-36 %, including lack of maturation and dominated by stenosis and thrombosis.

Local anesthesia associated with sedation is a validated method of anesthesia for made arteriovenous fistula but does not cause the motor block and not blocking vasospasm, deleterious to the surgery. Multiple injections necessary to cover the operating zone expose patient to pain and to intravascular injection of local anesthetics.

Regional anesthesia provides better conditions for realize more distal fistula. Sympathetic block provides arterial, venous vasodilation and decreases the incidence of vasospasm . It enables an increased flow rate at an early time fistula and faster maturation.

However, studies included low numbers of patient or are non-randomized. They cannot concluded a significant difference in the complication rate of arteriovenous fistula at an early time depending on the type of anesthesia .

This study aims to demonstrate that axillary block for surgical creation of arteriovenous fistula allows a reduction of complications at 6 weeks compared to local anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stade 4 or 5
* First creation of arteriovenous fistula on the side of the surgery
* written consent
* Health care system adherent
* No decision of juridical protection

Exclusion Criteria:

* Pregnancy or breast-feeding
* Participation to an other research study that may interfere with this study
* Brachial arterio-venous fistula creation (upper elbow crease)
* Antecedent of homolateral arteriovenous fistula (controlateral fistula non excluded)
* Other surgery on arteriovenous fistula (superficialisation procedure, refection…)
* Contraindications to local anesthetics : Ropivacaine or Lidocaine allergy
* Contraindication to regional anesthesia : homolateral axillary lymphadenectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-03; Primary Completion 2018-01-26 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Rate of early complications related to arteriovenous fistula regardless of type | 6 weeks after surgery
  Early complications include stenosis of arteriovenous fistula, thrombosis, lack of maturation, high flow, clinical steal syndrome, arteriovenous fistula infection, arteriovenous fistula hemorrhage, necessity of radiologic ou surgical reintervention,

SECONDARY OUTCOMES:
Rate of complications related to arteriovenous fistula regardless of type | 3 months after surgery
  Complications included stenosis of arteriovenous fistula, thrombosis, lack of maturation, high flow, clinical steal syndrome, arteriovenous fistula infection, arteriovenous fistula hemorrhage, necessity of radiologic ou surgical reintervention.
Rate of stenosis of arteriovenous fistula | 6 weeks after surgery
  stenosis of arteriovenous fistula : resistance index > 0.6, or peak velocity > 300 cm/s and residual diameter <3 mm
rate of thrombosis | 6 weeks after surgery
  thrombosis: resistance index = 1
incidence of abnormal arteriovenous fistula rate | 6 weeks after surgery
  abnormal arteriovenous fistula rate : lack of maturation (blood flow < 600 ml/min) or high flow (clinical heart failure, blood flow > 1200 ml/min)
incidence of clinical steal syndrome | 6 weeks after surgery
  clinical steal syndrome : trophic or neurological disorders
incidence of arteriovenous fistula infection | 6 weeks after surgery
incidence of arteriovenous fistula hemorrhage | 6 weeks after surgery
  arteriovenous fistula hemorrhage : spontaneous bleeding, post-puncture bleeding
necessity of radiologic ou surgical reintervention | 6 weeks after surgery
Rate of stenosis of arteriovenous fistula | 3 months after surgery
  stenosis of arteriovenous fistula : resistance index > 0.6, or peak velocity > 300 cm/s and residual diameter <3 mm
rate of thrombosis | 3 months after surgery
  thrombosis: resistance index = 1
incidence of abnormal arteriovenous fistula rate | 3 months after surgery
  abnormal arteriovenous fistula rate : lack of maturation (blood flow < 600 ml/min) or high flow (clinical heart failure, blood flow > 1200 ml/min)
incidence of clinical steal syndrome | 3 months after surgery
  clinical steal syndrome : trophic or neurological disorders
incidence of arteriovenous fistula infection | 3 months after surgery
incidence of arteriovenous fistula hemorrhage | 3 months after surgery
  arteriovenous fistula hemorrhage : spontaneous bleeding, post-puncture bleeding
necessity of radiologic ou surgical reintervention | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Thomas RIMMELE, MD, PhD, Principal Investigator — Hopital Edouard Herriot, Hospices Civils de Lyon, France
Locations (1):
- Hopital Edouard Herriot - Service Anesthésie et Réanimation, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Recommended by the KDOQI vascular access guidelines, antebrachial arteriovenous fistula is the best primary vascular access for hemodialysis in patients with end stage renal disease. The primary complications are common, of the order of 10-36 %, including lack of maturation and dominated by stenosis and thrombosis.~Local anesthesia associated with sedation is a validated method of anesthesia for made arteriovenous fistula but does not cause the motor block and not blocking vasospasm, deleterious to the surgery. Multiple injections necessary to cover the operating zone expose patient to pain and to intravascular injection of local anesthetics.~Regional anesthesia provides better conditions for realize more distal fistula. Sympathetic block provides arterial, venous vasodilation and decreases the incidence of vasospasm . It enables an increased flow rate at an early time fistula and faster maturation.~However, studies included low numbers of patient or are non-randomized. They cannot concluded a significant difference in the complication rate of arteriovenous fistula at an early time depending on the type of anesthesia .~This study aims to demonstrate that axillary block for surgical creation of arteriovenous fistula allows a reduction of complications at 6 weeks compared to local anesthesia